CLINICAL TRIAL: NCT02289443
Title: Comparison of Two Different Procedures Fabrication of Conventional Complete Dentures: a 10-year Follow-up Study of a Randomized Clinical Trial
Brief Title: a 10-year Follow-up Study of a Randomized Clinical Trial
Status: Completed | Type: Observational
Sponsor: Nihon University (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Yasuhiko Kawai, Professor, Nihon University
Other Study IDs: A09-E71-12B
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Edentulous
Keywords: complete dentures; 10-year follow-up; patient report outcomes
MeSH Terms: conditions — Mouth, Edentulous | interventions — Denture, Complete

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Simplified: Complete denture fabricated by simple way than the textbook traditional method.
  Interventions: Other: complete denture
- Traditional: Complete denture fabricated by textbook discribed traditional method.
  Interventions: Other: complete denture

INTERVENTIONS:
Other: complete denture — Comparison of different procedures

SUMMARY:
In this study, the investigators propose a 10-year follow up study of participants in a randomized clinical trial to compare the oral health-related quality of life (OHRQoL), as well as general and related satisfaction of conventional complete dentures fabricated using two different procedures.

DETAILED DESCRIPTION:
Study design A 10-year follow-up study of a randomized controlled clinical trial (RCT) carried out from 2001 to 2003, including assessment of patient satisfaction, denture repair/replacement and OHRQoL. Data will be gathered through telephone interviews. Since the contacts were last used a decade ago, the phone number may have been changed, but we will make every effort to find new numbers for any participant those contact information is no longer valid .

Subjects Patients who participated and completed 6-month follow-ups in the RCT (T group: 50, and S group: 54; total 104 subjects) will be contacted by telephone.

Interviews and blinding Potential subjects will be told that we are investigating conditions of their dentures 10-years after the delivery and that we will ask general questions, as well as for their ratings of satisfaction and OHRQoL regarding their dentures. After this, the subjects will be asked whether they are willing to respond to the interviews. If they agree, the interviewer will ask the questions according to a flow chart (Appendix 1a, b). The subjects will not be told to which group they had been assigned, and a blinded research assistant will carry out the interviews and data gathering. The research assistant worked with these participants during the active study 10 years before. Patients will be excluded if they cannot respond properly to the questions.

Questionnaires Data will be gathered by four questionnaires: socio-demographic (Q1: Appendix 2), denture history/oral health (Q2: Appendix 3), general and related satisfaction outcomes by answering VAS (visual analog scale) scores out of 100 (Q3: Appendix 4), and OHQOL measures (OHIP-EDENT) 12, 13 (Q4: Appendix 5).

Analysis Denture history The difference in number of people who keep and use the dentures at 10 years will be calculated in percentages. A Chi-squared test will be employed for the statistical analyses. Finally, the prevalence of problems associated with the dentures will be calculated.

Satisfaction The differences between the treatment groups in their general satisfaction ratings on 100mm VAS after the prostheses are worn for 10 years. A two-sample independent t-test will be employed. VAS items of comfort, stability, esthetics, retention, function and ease of cleaning are also included. These will be compared between the groups using t-tests.

OHRQoL OHIP-EDENT consists of 19 statements and responses varying from 0 to 4 on a Likert scale. The possible range between 0 and 76 will be derived individually and compared between the two groups. A two-sample independent t-test will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Who can be contact with telephone call and accept the interview

Exclusion Criteria:

* The line is closed, no response, who have deceased.
* Refused to answer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who participated and completed 6-month follow-ups in the RCT (T group: 50, and S group: 54; total 104 subjects) will be contacted by telephone.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 10years

SECONDARY OUTCOMES:
Denture repair/replacement | 10years
Oral Health related Quality of Life | 10years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kawai Y, Murakami H, Takanashi Y, Lund JP, Feine JS. Efficient resource use in simplified complete denture fabrication. J Prosthodont. 2010 Oct;19(7):512-6. doi: 10.1111/j.1532-849X.2010.00628.x. Epub 2010 Aug 16. PMID 20723019
- [Result] Kawai Y, Murakami H, Shariati B, Klemetti E, Blomfield JV, Billette L, Lund JP, Feine JS. Do traditional techniques produce better conventional complete dentures than simplified techniques? J Dent. 2005 Sep;33(8):659-68. doi: 10.1016/j.jdent.2005.01.005. PMID 16139697
- [Derived] Kawai Y, Muarakami H, Feine JS. Do traditional techniques produce better conventional complete dentures than simplified techniques? A 10-year follow-up of a randomized clinical trial. J Dent. 2018 Jul;74:30-36. doi: 10.1016/j.jdent.2018.04.027. Epub 2018 May 22. PMID 29758255